CLINICAL TRIAL: NCT03409913
Title: Conventional FDG PET/CT Accurately Diagnoses Temporal Arteritis in Glucocorticoid-naïve GCA Patients: a Case-control Study
Brief Title: Diagnostic Accuracy of FDG PET/CT of Cranial Arteries in GCA
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: Cranial_GCA_PET
Record Dates: First submitted 2018-01-18; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Giant Cell Arteritis
Keywords: positron emissions tomography; diagnostic accuracy; case-control
MeSH Terms: conditions — Giant Cell Arteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GCA cases: In a cohort of patients suspected of GCA based on the following inclusion criteria were 1) age ≥50 years, 2) CRP>15mg/l or ESR>40mm/h, 3) either a) cranial symptoms, b) new-onset extremity claudication or c) weight loss >5 kilograms or fever>38oC for >3 weeks, patients with a clinical diagnosis of GCA is identified.
  Interventions: Radiation: FDG PET/CT
- controls: Age-(+/- 3 years) and sex-matched malignant melanoma (MM) patients who had a follow-up metastatic-disease-free FDG PET/CT ≥6 months after MM resection
  Interventions: Radiation: FDG PET/CT

INTERVENTIONS:
Radiation: FDG PET/CT — Conventional FDG PET/CT including head in order to asses cranial arteries.
  Other Names: Temporal artery biopsy; Vascular ultrasound; Inflammatory biomarkers

SUMMARY:
A case-control study to evaluate the diagnostic accuracy of FDG uptake in cranial arteries by FDG PET/CT in the diagnosis of giant cell arteritis.

DETAILED DESCRIPTION:
Although older studies argue that FDG PET/CT cannot demonstrate inflammation in cranial arteries, e.g. temporal and maxillary arteries, the resolution of modern PET systems may have improved, making a case for FDG PET/CT. FDG PET/CT is increasingly used in giant cell arteritis (GCA) diagnosis due to its excellent diagnostic accuracy considering large-vessel involvement. In case of uncommon distribution of vessel involvement or marginally increased large-vessel FDG uptake, FDG PET/CT-specificity may be compromised. Hence, recognising FDG uptake in cranial arteries potentially adds to FDG PET/CTs diagnostic accuracy.

Objectives To evaluate the diagnostic accuracy of conventional FDG PET/CT of the cranial arteries in the diagnosis of GCA.

Methods In a cohort of consecutively included glucocorticoid-naïve patients suspected of new-onset GCA, patients with a clinical GCA diagnosis will be identified. Conventional FDG PET/CT and vascular ultrasound(US) was performed before treatment. Patients were referred for a temporal artery biopsy (TAB).

Controls are age-(+/- 3 years) and sex-matched malignant melanoma (MM) patients who had a follow-up metastatic-disease-free FDG PET/CT ≥6 months after MM resection.

Images will be assessed by 5 nuclear medicine physicians blinded to clinical symptoms and findings. Temporal (TA), maxillary (MA) and vertebral (VA) arteries will be visually assessed. Arterial FDG uptake more than FDG uptake in surrounding tissue is considered positive. Sensitivity, specificity and interreader agreement will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

Cases:

* 1) age ≥50 years, 2) CRP>15mg/l or ESR>40mm/h, 3) either a) cranial symptoms, b) new-onset extremity claudication or c) weight loss >5 kilograms or fever>38oC for >3 weeks and a clinical diagnosis of giant cell arteritis judged by expert rheumatologist.

Controls:

* age-(+/-3 years) and sex-matched malignant melanoma (MM) patients
* follow-up metastatic-disease-free FDG PET/CT ≥6 months after MM resection

Exclusion Criteria:

* Previous diagnosis of polymyalgia or giant cell arteritis
* immunosuppresive treatment within last month

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are sampled from tertiary hospital. Cases are identified in an established cohort of patients suspected og GCA in whom clinical assessment, including imaging procedures were performed before treatment.
  Controls are sampled among malignant melanoma patients who had a clinically indicated follow-up FDG PET/CT to evaluate disease freedom/progression.
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-10-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
PET positivity | Time of diagnosis/pre-treatment (cases)
  Presence of FDG uptake in temporal, maxillary and/or vertebral arteries assessed in order to evaluate sensitivity and specificity of PET of cranial arteries in the diagnosis of GCA

SECONDARY OUTCOMES:
Full-fillment of ACR criteria | Time of diagnosis
  PET sensitivity and specificity in the subpopulation of GCA patients full filling ACR criteria
Temporal artery biopsy | Time of diagnosis
  Correlation between temporal artery biopsy result and temporal artery FDG uptake
Temporal artery ultrasound | Time of diagnosis
  Correlation between temporal artery ultrasound result and temporal artery FDG uptake

CONTACTS AND LOCATIONS:
Overall Officials: Lars Christian Gormsen, MD, PhD, Study Chair — Department of Nuclear Medicine and PET centre, Aarhus University Hospital
Locations (1):
- Department of Rheumatology, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided